CLINICAL TRIAL: NCT06678789
Title: Evaluation of Low and High Nicotine Tobacco Free Nicotine Pouches as a Harm Reducing Substitute for Combustible Cigarettes - (Pack2Pouch)
Brief Title: Evaluation of Low and High Nicotine Tobacco Free Nicotine Pouches
Acronym: Pack2Pouch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00139710; 5K12DA031794 (NIH)
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cigarette Smoking; Nicotine Dependence; Smoking Cessation
Keywords: Smoking
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Nicotine (Experimental): High dosage nicotine pouches (6mg)
  Interventions: Behavioral: High Nicotine Dose
- Low Nicotine (Experimental): Low dosage nicotine pouches (3mg)
  Interventions: Behavioral: Low Nicotine Dose

INTERVENTIONS:
Behavioral: High Nicotine Dose — Will receive a 5-week supply of 6 mg Zyn pouches. Those who smoke 5-20 cigarettes per day will receive 1 tin per day = 35 tins, whereas those who smoke more will receive 2 tins/day [70 tins])
  Arms: High Nicotine
Behavioral: Low Nicotine Dose — Will receive a 5-week supply of 3 mg Zyn pouches. Those who smoke 5-20 cigarettes per day will receive 1 tin per day = 35 tins, whereas those who smoke more will receive 2 tins/day [70 tins])
  Arms: Low Nicotine

SUMMARY:
Tobacco-free oral nicotine pouches (such as Zyn brand) are a less harmful alternative to cigarette smoking. Pouches, however, contain nicotine, and addictive substance that is not risk-free. The present study is evaluating how well nicotine pouches, at different nicotine levels, help people switch away from smoking cigarettes. People who smoke cigarettes will be asked to answer questions about their tobacco product use and provide breath samples and cheek swab samples at an in-person visit to MUSC Charleston. Participants will then be provided with a 28-day supply of nicotine pouches, and will be asked to switch from smoking to pouches over the course of 4 weeks. Finally, participants will complete a final visit at MUSC, and will answer more questions about their tobacco use 1-month later.

DETAILED DESCRIPTION:
The proposed research project evaluates the potential for tobacco-free oral nicotine pouches (TFNPs) to serve as harm reduction tools at two nicotine concentrations, inclusive of behavioral and biomarker outcomes, using a clinical trial design. Specifically, in a randomized pilot study, participants who smoke will be recruited and sent TFNPs to sample for 4 weeks in either high (6 mg) or low (3 mg) nicotine content strengths. Participants will report tobacco use behaviors and submit biological samples throughout the study. This design allows for evaluation of the effect of nicotine content within alternative, harm-reducing tobacco products on key outcomes including: 1) complete switching from cigarette smoking to non-cigarette product use; 2) cigarette smoking reduction; 3) changes in biomarkers of harm (DNA damage, respiratory symptoms), 4) nicotine dependence, and 5) subjective effects of product use.

ELIGIBILITY:
Inclusion Criteria:

* Age 21+
* current cigarette smoking (25+ days per previous month, 5 or more cigarettes/day, for greater than 1yr, greater than 100 lifetime cigarettes)
* have not used TNFPs more than 5 times during their lifetime
* willing and able to attend 2 in-person visits in Charleston (to assess biomarkers)
* have internet access

Exclusion Criteria:

* Lack of proficiency in English.
* Use of other combustible tobacco products (i.e., cigars, cigarillos, hookahs) and/or other non-combusted nicotine/tobacco products (i.e., e-cigarettes, smokeless tobacco) in the past 30 days.
* Current use of smoking cessation medications (i.e., varenicline, bupropion, nicotine replacement therapy).
* Use of marijuana within the past month, and unwillingness to abstain from marijuana during course of study.
* Medical conditions contraindicated to NRT use (including pregnancy, breastfeeding, and nursing, past month myocardial infarction, current untreated cardiac arrhythmia, current severe angina, current uncontrolled severe vascular disease).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Switching | Day 28 and Day 56
  Switching will be defined at 7-day point-prevalence biochemically-confirmed abstinence from cigarettes alongside self-reported use of nicotine pouches. Non-responders and missing data will be coded as smoking.
Smoking Reduction | Day 28 and Day 56
  Baseline and daily survey data will be used to calculate the change of smoking (average cigarettes per day) between groups from baseline to end of sampling.

SECONDARY OUTCOMES:
Tobacco-Free Oral Nicotine Pouches (TFNP) Use | Day 28
  Daily surveys will capture number of days of TFNP use, regardless of smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Palmer, PhD., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified self-report data and outcomes from biosample analyses will be shared upon reasonable request. Biological samples will not be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data and supporting information will be shared 1 year after study results are published.
Access Criteria: Academic researchers who are not affiliated with or funded by the tobacco industry (including their consultants and non-profit organizations) may request access.